CLINICAL TRIAL: NCT00042120
Title: Pesticides and Risk in the Agricultural Health Study
Brief Title: Farming and Movement Evaluation Study (FAME)
Acronym: FAME
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Caroline M. Tanner, MD, Ph.D., The Parkinson's Institute
Other Study IDs: 10803-CP-001; NCT00342914 (obsolete NCT alias)
Record Dates: First submitted 2002-07-24; First posted 2002-07-26 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2009-08

CONDITIONS: Parkinson's Disease; Movement Disorders
Keywords: Parkinson's disease; Movement Disorders; Epidemiological Study
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
The long term goal of this research is to elucidate the cause(s) of Parkinson's disease, with a focus on environmental determinants. We propose to investigate the relationship between Parkinson's disease and exposure to pesticides and other factors by conducting a nested case-control study in the Agricultural Health Study.

DETAILED DESCRIPTION:
The long term goal of this research is to elucidate the cause(s) of Parkinson's disease, with a focus on environmental determinants. We propose to investigate the relationship between Parkinson's disease and exposure to pesticides and other factors by conducting a nested case-control study in the Agricultural Health Study.

The Agricultural Health Study is a cohort study of 52,000 licensed pesticide applicators and 32,000 of their spouses, conducted in North Carolina and Iowa. It is a joint effort of the National Cancer Institute, the National Institute of Environmental Health Sciences, and the US Environmental Protection Agency.

The studies proposed here take full advantage of the Agricultural Health Study. We believe that this work could provide a critical and dramatic next step in furthering our knowledge of environmental determinants of PD, and thereby take us closer to our goal of finding its cause(s)

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited from members of the Agricultural Health Study cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2001-04; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Tanner, Principal Investigator — The Parkinson's Institute
Locations (1):
- The Parkinson's Institute, Sunnyvale, California, United States